CLINICAL TRIAL: NCT03565120
Title: The Efficacy and Toxicity of Aggressive Thoracic Radiotherapy for Stage Ⅳ Non-Small Cell Lung Cancer Patients With Controlled Extrathoracic Disease
Brief Title: Aggressive Thoracic Radiotherapy for Stage Ⅳ Non Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: yu gengsheng (Other)
Responsible Party: Sponsor-Investigator, yu gengsheng, Vice director of Oncology department, Jiangmen Central Hospital
Organization: Jiangmen Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATR-NSCLC
Record Dates: First submitted 2018-05-21; First posted 2018-06-21 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Stage IV; Thoracic Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm-R (Experimental): patients in this arm will receive aggressive thoracic radiotherapy.
  Interventions: Radiation: Aggressive Thoracic Radiotherapy

INTERVENTIONS:
Radiation: Aggressive Thoracic Radiotherapy — The target of the radiotherapy includes primary tumor and the locoregional positive lymph nodes, with a dose(BED)≥53Gray(Gy)

SUMMARY:
This phase II trial studies the safety and efficacy of aggressive thoracic radiotherapy in treating patients with non-small cell lung cancer that has not progressed after the first line systemic therapy. In this trial, patients with stage Ⅳ non small cell lung cancer who did not progress after first line systemic therapy will receive the aggressive thoracic radiotherapy, and the safety and efficacy of aggressive thoracic radiotherapy will be evaluated. The primary end points of the study are overall survival (OS), the secondary end points are local control rate, local progression free survival(LPFS), PFS, and toxicity and quality of life(QOL).

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed NSCLC
* stage IV disease
* no progression after first line systemic therapy
* 18 to 80 years of age
* Karnofsky performance status(KPS) score ≥70%
* no contraindications to radiation therapy
* presumed ability to tolerate thoracic radiation therapy to a BED≥53Gy

Exclusion Criteria:

* a history of thoracic surgery, radiation therapy, or more than first line chemotherapy
* pregnancy or lactation at the time of enrollment
* previous malignancy or other concomitant malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
OS | two years after the beginning of first line systemic therapy
  overall survival

SECONDARY OUTCOMES:
LPFS | 1 year after the beginning of first line systemic therapy
  local progression free survival
PFS | 1 year after the beginning of first line systemic therapy
  progression free survival
toxicity related to the radiotherapy | from the beginning of radiotherapy to the 3 month after the completion of radiotherapy
  assess according to the National Cancer Institute-Common Terminology Criteria for Adverse Events 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Yu Gengsheng, master, Study Director — jiangmen cenctral hospital
Locations (1):
- Jiangmen central hospital, Jiangmen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kepka L, Olszyna-Serementa M. Palliative thoracic radiotherapy for lung cancer. Expert Rev Anticancer Ther. 2010 Apr;10(4):559-69. doi: 10.1586/era.10.22. PMID 20397921
- [Background] Fairchild A, Harris K, Barnes E, Wong R, Lutz S, Bezjak A, Cheung P, Chow E. Palliative thoracic radiotherapy for lung cancer: a systematic review. J Clin Oncol. 2008 Aug 20;26(24):4001-11. doi: 10.1200/JCO.2007.15.3312. PMID 18711191
- [Background] Koshy M, Malik R, Mahmood U, Rusthoven CG, Sher DJ. Comparative effectiveness of aggressive thoracic radiation therapy and concurrent chemoradiation therapy in metastatic lung cancer. Pract Radiat Oncol. 2015 Nov-Dec;5(6):374-82. doi: 10.1016/j.prro.2015.07.009. Epub 2015 Aug 1. PMID 26412340
- [Background] Flannery TW, Suntharalingam M, Regine WF, Chin LS, Krasna MJ, Shehata MK, Edelman MJ, Kremer M, Patchell RA, Kwok Y. Long-term survival in patients with synchronous, solitary brain metastasis from non-small-cell lung cancer treated with radiosurgery. Int J Radiat Oncol Biol Phys. 2008 Sep 1;72(1):19-23. doi: 10.1016/j.ijrobp.2007.12.031. Epub 2008 Feb 14. PMID 18280058
- [Background] Su SF, Hu YX, Ouyang WW, Lu B, Ma Z, Li QS, Li HQ, Geng YC. Overall survival and toxicities regarding thoracic three-dimensional radiotherapy with concurrent chemotherapy for stage IV non-small cell lung cancer: results of a prospective single-center study. BMC Cancer. 2013 Oct 12;13:474. doi: 10.1186/1471-2407-13-474. PMID 24118842
- [Background] Sheu T, Heymach JV, Swisher SG, Rao G, Weinberg JS, Mehran R, McAleer MF, Liao Z, Aloia TA, Gomez DR. Propensity score-matched analysis of comprehensive local therapy for oligometastatic non-small cell lung cancer that did not progress after front-line chemotherapy. Int J Radiat Oncol Biol Phys. 2014 Nov 15;90(4):850-7. doi: 10.1016/j.ijrobp.2014.07.012. Epub 2014 Sep 9. PMID 25216859
- [Background] Chiang Y, Yang JC, Hsu FM, Chen YH, Shih JY, Lin ZZ, Lan KH, Cheng AL, Kuo SH. The Response, Outcome and Toxicity of Aggressive Palliative Thoracic Radiotherapy for Metastatic Non-Small Cell Lung Cancer Patients with Controlled Extrathoracic Diseases. PLoS One. 2015 Dec 31;10(12):e0145936. doi: 10.1371/journal.pone.0145936. eCollection 2015. PMID 26720170
- [Background] Wang J, Ji Z, Wang X, Liang J, Hui Z, Lv J, Zhou Z, Yin W, Wang L. Radical thoracic radiotherapy may provide favorable outcomes for stage IV non-small cell lung cancer. Thorac Cancer. 2016 Mar;7(2):182-9. doi: 10.1111/1759-7714.12305. Epub 2015 Sep 13. PMID 27042220
- [Background] Su S, Hu Y, Ouyang W, Ma Z, Li Q, Li H, Wang Y, Wang X, Li T, Li J, Chen M, Lu Y, Bai Y, He Z, Lu B. Might radiation therapy in addition to chemotherapy improve overall survival of patients with non-oligometastatic Stage IV non-small cell lung cancer?: Secondary analysis of two prospective studies. BMC Cancer. 2016 Nov 21;16(1):908. doi: 10.1186/s12885-016-2952-3. PMID 27871270